CLINICAL TRIAL: NCT01963533
Title: The Roles of Age, Comorbidity, and Telomere Length in Lung Cancer Treatment and Prognosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201207006RIC
Record Dates: First submitted 2013-10-08; First posted 2013-10-16 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-10

CONDITIONS: Lung Cancer
Keywords: lung cancer; telomere length; comorbidity; Eastern Cooperation Oncology Group (ECOG); chemotherapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators hypothesize that the age-adjusted telomere length in lung cancer patients before chemotherapy may be correlated to comorbidity status and predict outcome. The change of telomere length shortening after chemotherapy may relate to treatment side effect and treatment response.

DETAILED DESCRIPTION:
Except chemotherapy, telomere shortening were also related to a variety of cellular stress, including hydrogen peroxide, UV, and x-irradiation, transforming growth factor-beta, overexpression of oncogenes such as Ha-Ras. The cellular stress induced telomere shortening and/or telomere dysfunction and promote accelerated senescence in normal and malignant cells. Oxidative stress, which presented in several chronic inflammatory diseases, such as atherosclerosis, coronary artery disease, and chronic obstructive airway disease, was also found to be correlated with telomere shortening.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are newly diagnosed as lung cancer and prepared for scheduled chemotherapy.
2. The diagnosis is based on pathology via surgical specimen, or biopsy; or cytology via lung, lymph node aspiration or effusion study.

Exclusion criteria:

includes clinical diagnosis of lung cancer without pathology or cytology proving, combined with other type malignancy, and expected short survival time less than one month.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are newly diagnosed as lung cancer and prepared for scheduled chemotherapy in National Taiwan University Hospital will be enrolled for screening. The diagnosis is based on pathology via surgical specimen, or biopsy; or cytology via lung, lymph node aspiration or effusion study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The correlation between telomere length shortening and cancer treatment outcome | 5 years
  The clinical data, including age, gender, clinical presentation, performance status, disease stage at diagnosis, initial treatment modality, progression-free survival of initial treatment, and survival duration will be recorded. Blood sample collection, quality of life, and cognitive function assessment will be performed before chemotherapy, one and four weeks after initial chemotherapy for telomere length measurement. Telomere length is measured by quantitative polymerase chain reaction(qPCR). Patients' characteristics are compared with chi-square test. Progression-free survival and survival time are analyzed by Kaplan-Meier with log rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Yu Chen, PhD, Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan